CLINICAL TRIAL: NCT01037777
Title: Prospective Study of Individuals at Risk for Spinocerebellar Ataxia Type 1, Type 2, Type 3, Type 6 and Type 7 (SCA1, SCA2, SCA3, SCA6, SCA7)
Brief Title: RISCA : Prospective Study of Individuals at Risk for SCA1, SCA2, SCA3, SCA6, SCA7
Acronym: RISCA
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C08-37
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Spinocerebellar Ataxias
Keywords: individuals at risk for SCA1, SCA2, SCA3, SCA6 and SCA7
MeSH Terms: conditions — Spinocerebellar Ataxias

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective

GROUPS / COHORTS (2):
- presymptomatic carriers
- non carrier relatives

SUMMARY:
The spinocerebellar ataxias (SCAs) are a clinically and genetically heterogeneous group of autosomal dominantly inherited progressive ataxia disorders. It is estimated that there are 30,000 individuals in the European Community that directly descend from individuals affected by a SCA disorder and thus carry a 50% risk of having inherited an SCA mutation. These at risk individuals provide a unique research opportunity to prospectively study the presymptomatic phase of SCA disorders and to identify the earliest and most sensitive clinical signs and biological markers that herald the onset of the illness. This information is of critical importance for the development of future therapeutic interventions aimed at postponing the clinical onset of ataxia.

We therefore propose to perform a prospective observational study of individuals at risk for the most common SCA disorders, SCA1, SCA2, SCA3 and SCA6 (RISCA). It is our aim to answer the following questions: (1) What is the incidence of disease manifestation in mutation carriers? (2) Which clinical signs precede the onset of manifest ataxia in SCA1, SCA2, SCA3 and SCA6? (3) What are the prevalence and incidence of preceding signs? (4) Are the prevalence and incidence of preceding signs affected by genotype, gender, age, estimated time until disease manifestation and repeat length? (5) Does the presence of certain preceding signs predict the manifestation of ataxia ? (6) Are there MRI alterations that precede the onset of ataxia? It is planned to enroll 480 study participants and to follow them at regular intervals over six years. At each visit, study participants are asked in a structured interview for a number of predefined clinical signs that potentially precede the onset of ataxia. In addition, the following self-assessment scales will be applied: Pittsburgh Sleep Quality Index (PSQI), Diagnostic Criteria for Restless Legs Syndrome, Patient´s Health Questionnaire (PHQ-9). All study participants will undergo a physical examination including the Scale for the Assessment and Rating of Ataxia (SARA). Study participants will further perform the SCA Functional Composite (SCA-FC) which is a comprehensive measure of functional capacity based on results in quantitative tests related to gait (8m timed walk), speech (PATA rate) and hand function (9 hole pegboard). In a subset of study participants, we will record eye movements and obtain volumetric MRIs. The study will also be used to collect and store blood and urine samples for proteomic and gene expression studies.

RISCA is conducted by the Ataxia Study Group (ASG). It relies on the network structure created by the EUROSCA project.

ELIGIBILITY:
Inclusion Criteria:

* individuals at risk for spinocerebellar ataxia type 1, type 2, type 3, type 6 and type 7 (SCA1, SCA2, SCA3, SCA6 and SCA7)
* age between 18 and 50 years old for SCA1, SCA2, SCA3 or SCA7
* age between 35 and 70 years old for SCA6
* no clinical sign of ataxia (SARA < 3)

Exclusion Criteria:

* no writing consent
* no family members affected
* presence of clinical sign of ataxia (SARA > 3)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French population
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2009-05-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pitié Salpêtrière Hospital, Paris, France

REFERENCES:
- [Derived] Wilke C, Mengel D, Schols L, Hengel H, Rakowicz M, Klockgether T, Durr A, Filla A, Melegh B, Schule R, Reetz K, Jacobi H, Synofzik M. Levels of Neurofilament Light at the Preataxic and Ataxic Stages of Spinocerebellar Ataxia Type 1. Neurology. 2022 May 17;98(20):e1985-e1996. doi: 10.1212/WNL.0000000000200257. Epub 2022 Mar 9. PMID 35264424
- [Derived] Jacobi H, du Montcel ST, Romanzetti S, Harmuth F, Mariotti C, Nanetti L, Rakowicz M, Makowicz G, Durr A, Monin ML, Filla A, Roca A, Schols L, Hengel H, Infante J, Kang JS, Timmann D, Casali C, Masciullo M, Baliko L, Melegh B, Nachbauer W, Burk-Gergs K, Schulz JB, Riess O, Reetz K, Klockgether T. Conversion of individuals at risk for spinocerebellar ataxia types 1, 2, 3, and 6 to manifest ataxia (RISCA): a longitudinal cohort study. Lancet Neurol. 2020 Sep;19(9):738-747. doi: 10.1016/S1474-4422(20)30235-0. PMID 32822634
- [Derived] Tezenas du Montcel S, Durr A, Rakowicz M, Nanetti L, Charles P, Sulek A, Mariotti C, Rola R, Schols L, Bauer P, Dufaure-Gare I, Jacobi H, Forlani S, Schmitz-Hubsch T, Filla A, Timmann D, van de Warrenburg BP, Marelli C, Kang JS, Giunti P, Cook A, Baliko L, Melegh B, Boesch S, Szymanski S, Berciano J, Infante J, Buerk K, Masciullo M, Di Fabio R, Depondt C, Ratka S, Stevanin G, Klockgether T, Brice A, Golmard JL. Prediction of the age at onset in spinocerebellar ataxia type 1, 2, 3 and 6. J Med Genet. 2014 Jul;51(7):479-86. doi: 10.1136/jmedgenet-2013-102200. Epub 2014 Apr 29. PMID 24780882
- [Derived] Jacobi H, Reetz K, du Montcel ST, Bauer P, Mariotti C, Nanetti L, Rakowicz M, Sulek A, Durr A, Charles P, Filla A, Antenora A, Schols L, Schicks J, Infante J, Kang JS, Timmann D, Di Fabio R, Masciullo M, Baliko L, Melegh B, Boesch S, Burk K, Peltz A, Schulz JB, Dufaure-Gare I, Klockgether T. Biological and clinical characteristics of individuals at risk for spinocerebellar ataxia types 1, 2, 3, and 6 in the longitudinal RISCA study: analysis of baseline data. Lancet Neurol. 2013 Jul;12(7):650-8. doi: 10.1016/S1474-4422(13)70104-2. Epub 2013 May 22. PMID 23707147